CLINICAL TRIAL: NCT01308216
Title: Efficacy of Transcranial Laser Therapy for Improving Upper Extremity Functional Recovery in Hemiplegic Patients From Ischemic Stroke
Brief Title: Transcranial Laser Therapy in the Rehabilitation of Hemiplegic Patients From Ischemic Stroke
Acronym: REHELA
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Based in the negative of patients to shave de hair.
Sponsor: Hospital Universitario Ramon y Cajal (Other)
Responsible Party: Principal Investigator, RAMON MONTES MOLINA, Physical Therapy, Hospital Universitario Ramon y Cajal
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RyC-10
Record Dates: First submitted 2011-03-03; First posted 2011-03-04 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2011-11

CONDITIONS: Hemiplegia
Keywords: Transcranial Laser Therapy; Hemiplegia; Rehabilitation; Physiotherapy; Ischemic stroke
MeSH Terms: conditions — Hemiplegia; Ischemic Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Transcranial low level laser therapy (Experimental): Transcranial laser therapy is applied by automatic scanning over both hemispheres and the patients undergoing also a standard rehabilitation program based on therapeutic exercises.
  Interventions: Procedure: low level laser therapy procedure
- Control (Active Comparator): The patients undergoing only a standard rehabilitation program based on therapeutic exercises.
  Interventions: Procedure: low level laser therapy procedure

INTERVENTIONS:
Procedure: low level laser therapy procedure — Transcranial low level laser therapy by automatic scanning noncontact over both cerebral hemispheres.
  Other Names: COMBY 3 Terza Serie C-LASER; ASA.

SUMMARY:
The aim of this study is to determine the efficacy of transcranial laser therapy applied in automatic noncontact scanning mode for improving functional disability in patients with hemiplegia from ischemic stroke undergoing a rehabilitation program.

DETAILED DESCRIPTION:
Transcranial laser therapy is applied with an InGa(Al)As diode laser.The laser in automatic scanning is applied over both cerebral hemisphere during 15 sessions. Patients simultaneously performed a program of therapeutic exercises 3 days a week. Outcome measures were the Fugl-Meyer Upper Extremity scale, which assessed upper limb motor function, and the Barthel index, which assessed general functional disability.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with hemiplegia secondary to cerebral stroke ischemic.
2. Requirement of shaving the scalp area.
3. Initiation of the TLT procedure begins between 70 and 100 days after stroke onset.
4. Informed written consent before enrolling in the study.

Exclusion Criteria:

1. Hemiplegia secondary to hemorrhagic stroke.
2. Metallic brain implants.
3. Neurodegenerative disorders.
4. Bilateral motor problems.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2010-11; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Scale | 20 minutes
  The upper extremity Fugl-Meyer subscale (0-66) considers flexor and extensor synegies as well as reflex activity and coordination and is specific for grading motor impairments.

SECONDARY OUTCOMES:
Barthel index | 10 minutes
  Barthel index (0-100) is composed of 10 items and assesses activities related to clothing,nourishment,personal hygiene and transference.

CONTACTS AND LOCATIONS:
Overall Officials: Ramón Montes-Molina, PT, Principal Investigator — Hospital University Ramon y Cajal. IRYCIS.Madrid
Locations (1):
- Hospital Ramon y Cajal, Madrid, Madrid, Spain